CLINICAL TRIAL: NCT02727647
Title: Comparison of Different Prophylaxis Regimens for Moderate to Severe Hemophilia A Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Darintr Sosothikul, Associate professor, Chulalongkorn University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3125056
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2015-10

CONDITIONS: Hemophilia A
Keywords: Moderate hemophilia A; Severe hemophilia A; Intermediate dose prophylaxis; Low dose prophylaxis
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): FVIII concentration at 35-40 U/kg/dose 1 time/week for 5 months
  Interventions: Drug: FVIII
- Arm 2 (Experimental): FVIII concentration at 15-20 U/kg/dose 2 time/week for 5 months
  Interventions: Drug: FVIII

INTERVENTIONS:
Drug: FVIII — FVIII concentration 35-40 U/kg/dose 1 time/week for 5 months
  Other Names: Hemofil-M
  Arms: Arm 1
Drug: FVIII — FVIII concentration 15-20 U/kg/dose 1 time/week for 5 months
  Other Names: Hemofil-M
  Arms: Arm 2

SUMMARY:
Title: Comparison of different prophylaxis regimens for hemophilia A pediatric patients Principal Investigator: Assistant Professor Darintr Sosothikul, MD Research Question: Does different factor VIII dosage effect outcome of hemophilia treatment in term of breakthrough bleeding, number of hospital stay and day-off from school? Type Research: Clinical research

Study design: Single center clinical trials

Concise methodology:

1. Study Population: Children with hemophilia A who received treatment at KCMH from May 2015 to March 2016 will be enrolled in this study. The consent will be obtained before the study.
2. Observation and measurement:

   1. History, interesting clinical data and laboratory data will be recorded in Clinical record Form (CRF)
   2. Measurement:

   i. Complete blood count (CBC), Factor VIII level, Factor VIII inhibitor level ii. Number of breakthrough bleedings, number of hospital stay and day-off from school iii. Joint score from Hemophilia Joint Health Score 2.1 iv. EQ-5D-5L quality of life assessment score
3. Data analysis: The p-value of less than 0.05 will be considered statistically significant. Mann-Whitney test will be used to test correlation of these variables (CBC, Factor VIII level, Factor VIII inhibitor level, Number of breakthrough bleedings, number of hospital stay, day-off from school, Hemophilia Joint Health Score 2.1, EQ-5D-5L quality of life assessment score) Sample size: 16 patients

Potential impacts:

The outcomes of different factor VIII concentrate dose between 15-20 U/kg/dose 2 times/week and 35-40 U/kg/dose 1 time/week will be revealed. These outcomes include number of breakthrough bleeding, number of hospital stay, day-off from school, joint health and quality of life. The result of this study will guide further study on optimal dose and duration of factor VIII treatment of hemophilia A patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia patients with moderate (factor level 1-3%) or severe (factor level <1%) severity

Exclusion Criteria:

* Platelet count less than 100,000 /mm3 or other bleeding tendency
* Hemophilia patients who have FVIII inhibitor >0.6 BU (modified Nijmogen method)
* Hemophilia patients who have no bleeding symptoms

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Annualized bleeding rate per year | 10 months

SECONDARY OUTCOMES:
Hemophilia joint health score | 10 months
Amount of FVIII use | 10 months
Quality of life score | 10 months
  EQ-5D-5L (Thailand version)
Number of hospital stays | 10 months
Number of school days loss | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Darintr Sosothikul, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Division of Hemato/oncology, Department of Pediatrics, Faculty of medicine,Chulalongkorn U, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No